CLINICAL TRIAL: NCT06466889
Title: Genetic, Multiomic and Cytokine-based Mapping of Patients With Mastocytosis/Hypertryptasemia at the University Hospital of Zurich German: Mastozytose-Register: Datenerfassung Und Weiterverwendung Von Biologischem Material Von Patienten Mit Mastozytose, Welche am Universitätsspital Zürich Behandelt Werden
Brief Title: Mastocytosis Registry (of Zurich)
Acronym: MastoR
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2020-01568
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Mastocytosis; Hypertryptasemia
Keywords: mast cell disease
MeSH Terms: conditions — Mastocytosis; Mast Cell Activation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — PBMC, skin samples, gut tissue, bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mastocytosis: Diagnosed mastocytosis according to WHO criteria
- Hypertryptasemia: Repeated elevated serum tryptase with no underlying mastocytosis or no bone marrow biopsy performed

SUMMARY:
The study aims to summarize patients with mastocytosis and hypertryptasämia (without underlying mastocytosis or no bone marrow biopsy) in relation to demographic information, clinical progress and treatment courses. Biologic samples are collected from available routine diagnostics (serum, skin tissue, gut mucosa, bone marrow, and others) for further use in experimental research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with mastocytsis/hypertryptasemia which are treated at the university hospital of Zurich
* available informed consent

Exclusion Criteria:

* denied consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients with mastocytosis or hypertryptasemia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographics | 2010-2025
  In the registry we collect patient's demographic data e.g. age, gender, comorbidities, smoking, preexisting atopic disease and other to look for associations to mast cell diseases.
Disease progression | 2010-2025
  Patients will followed up over time to get more insight in disease progression.If there is progression detected (e.g. cutaneous mastocytosis to systemic mastocytosis or ISM to advanced forms) those cases will be carefully looked at to identify triggering factors and biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
set up multicenter registry, patient data will be anonymous